CLINICAL TRIAL: NCT01566604
Title: A 26-week Treatment, Randomised, Double-blind, Placebo-controlled, Parallel Group Study to Assess the Efficacy, Safety and Tolerability of NVA237 (50 µg o.d.) in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Efficacy, Safety and Tolerability of NVA237 in Patients With Chronic Obstructive Pulmonary Disease
Acronym: GLOW7
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CNVA237A2309
Record Dates: First submitted 2012-03-27; First posted 2012-03-29 (Estimated); Results first posted 2014-08-08 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-07

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Chronic obstructive pulmonary disease (COPD); NVA237
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Glycopyrrolate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- NVA237 (Experimental): NVA237 50 µg once daily delivered via a single dose dry powder inhaler
  Interventions: Drug: NVA237
- Placebo (Placebo Comparator): Placebo once daily delivered via a single dose dry powder inhaler
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NVA237 — Delivered via a single dose dry powder inhaler
  Arms: NVA237
Drug: Placebo — Delivered via a single dose dry powder inhaler
  Arms: Placebo

SUMMARY:
This study will assess of the efficacy and safety of a once-daily, 50µg inhalation of NVA237 in moderate to severe chronic obstructive pulmonary disease (COPD) patients over 26 weeks treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults aged ≥40 years, who have signed an Informed Consent Form prior to initiation of any study-related procedure
* With moderate to severe stable COPD (Stage II or Stage III).
* Current or ex-smokers who have a smoking history of at least 10 pack years (Ten pack- years are defined as 20 cigarettes a day for 10 years, or 10 cigarettes a day for 20 years).
* Post-bronchodilator FEV1 ≥30% and < 80% of the predicted normal, and post-bronchodilator FEV1/FVC < 0.7 at Visit 2 (Day -14) (post means: record FEV1 and FVC 45 min after administering ipratropium).
* Symptomatic patients, according to daily electronic diary data between Visit 2 (Day -14) and Visit 3 (Day 1), with a total score of 1 or more on at least 4 of the last 7 days prior to Visit 3

Exclusion Criteria:

* With a history of malignancy of any organ system (including lung cancer), treated or untreated, within the past 5 years whether or not there is evidence of local recurrence or metastases, with the exception of localized basal cell carcinoma of the skin.
* Patients with any history of asthma indicated by (but not limited to) a blood eosinophil count > 600/mm3 (at Visit 2) or onset of symptoms prior to age 40 years. Patients without asthma but who have a blood eosinophil count >600/mm3 at Visit 2 are excluded.
* Patients with concomitant pulmonary disease, e.g. pulmonary tuberculosis (unless confirmed by imaging to be no longer active) or clinically significant bronchiectasis, sarcoidosis and interstitial lung disorder.
* Patients with lung lobectomy or lung volume reduction or lung transplantation.
* Patients with known history and diagnosis of α-1 antitrypsin deficiency.
* Patients who have had a COPD exacerbation that required treatment with antibiotics, systemic steroids (oral or intravenous) or hospitalization in the 6 weeks prior to Visit 1 Patients who have had a respiratory tract infection within 6 weeks prior to Visit 1.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2012-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (26):
- China (16):
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Nanning, Guangxi
  - Novartis Investigative Site, Shijiazhuang, Hebei
  - Novartis Investigative Site, Changsha, Hunan
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Suzhou, Jiangsu
  - Novartis Investigative Site, Nanchang, Jiangxi
  - Novartis Investigative Site, Shengyang, Liaoning
  - Novartis Investigative Site, Shanghai, Shanghai Municipality
  - Novartis Investigative Site, Xi’an, Shanxi
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Chongqing
  - Novartis Investigative Site, Guangzhou
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Tianjin
- India (2):
  - Novartis Investigative Site, Dehli, New Delhi
  - Novartis Investigative Site, Coimbatore, Tamil Nadu
- Philippines (4):
  - Novartis Investigative Site, Bulacan, Philippines
  - Novartis Investigative Site, Manila, Philippines
  - Novartis Investigative Site, Las Piñas
  - Novartis Investigative Site, Quezon City
- South Korea (4):
  - Novartis Investigative Site, Seoul, Seoul
  - Novartis Investigative Site, Daejeon
  - Novartis Investigative Site, Incheon
  - Novartis Investigative Site, Seoul

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized in a 2: 1 ration to NVA237 and Placebo, respectively.
Period: Overall Study
Arm/Group | NVA237 | Placebo
Started | 306 | 154
Safety Set | 305 | 154
Full Analysis Set (FAS) | 305 | 154
FAS, Serial Spirometry Subgroup | 134 | 58
Completed | 282 | 143
Not Completed | 24 | 11
Not completed — Patient's inability to use the device | 1 | 0
Not completed — Administrative problems | 1 | 0
Not completed — Lack of Efficacy | 1 | 2
Not completed — Protocol deviation | 2 | 0
Not completed — Abnormal laboratory value | 2 | 0
Not completed — Death | 4 | 1
Not completed — Adverse Event | 4 | 2
Not completed — Withdrawal by Subject | 9 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NVA237 | Placebo | Total
Number analyzed (Participants) | 305 | 154 | 459
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.6 (7.84) | 65.0 (8.29) | 64.7 (7.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 294 | 145 | 439

OUTCOME MEASURES:

1. Primary Outcome: Trough Forced Expiratory Volume in One Second (FEV1)
Description: Baseline FEV1 was defined as the average of the -45 min and -15 min FEV1 values taken on day 1 prior to the first dose of study medication. Trough FEV1 was defined as the mean of the post-dose 23 h 15 min and the 23 h 45 min FEV1 values. FEV1 was measured using central spirometry according to ATS/ERS standardization. Trough FEV1 was analyzed using a MIXED model for the full analysis set population. The model contained treatment as a fixed effect with the baseline FEV1 measurement, FEV1 prior to inhalation of short acting bronchodilator, FEV1 45 min post inhalation of short acting bronchodilator and baseline inhaled corticosteroids (ICS) use as covariates.
Time Frame: 12 weeks
Population: The number of participants considered for the analysis was from the full analysis set (randomized participants who received at least one dose of study medication). However, participants analyzed had both baseline and week 12 values.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | NVA237 | Placebo
Number analyzed (Participants) | 296 | 147
Liters | 1.204 (0.0135) | 1.063 (0.0160)

2. Secondary Outcome: Transition Dyspnea Index (TDI) Score
Description: Dyspnea was measured at baseline using the Baseline Dyspnea Index (BDI) and during the treatment period using the TDI, which captures changes from baseline. The BDI and TDI each have three domains: functional impairment, magnitude of task and magnitude of effort, and each domain scored from -3 (major deterioration) to +3 (major improvement), giving an overall score of -9 to +9. A negative score indicates deterioration from baseline. A TDI focal score of 1 is considered to be a clinically significant improvement from baseline.
Time Frame: Baseline, week 12, week 26
Population: The number of participants considered for the analysis was from the full analysis set (randomized participants who received at least one dose of study medication). However, for a given time frame, analyzed participants had values at both baseline and the corresponding time frame, i.e. week 12 or week 26.
Measure: Least Squares Mean (Standard Error); unit: score
Arm/Group | NVA237 | Placebo
Number analyzed (Participants) | 305 | 154
score
  week 12 (n=288,141) | 2.8 (0.32) | 1.6 (0.34)
  week 26 (n=284,140) | 3.0 (0.31) | 2.0 (0.34)

3. Secondary Outcome: Change From Baseline in Daily Rescue Medication Use (Number of Puffs)
Description: The participant recorded the rescue medication taken in an electronic diary between visits and in the spirometry device during study visits. Daytime and nighttime rescue medication use (number of puffs) over 26 weeks was analyzed.
Time Frame: Baseline, 26 weeks
Population: Full Analysis Set: The full analysis set included all randomized participants who received at least one dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: Number of puffs
Arm/Group | NVA237 | Placebo
Number analyzed (Participants) | 305 | 154
Number of puffs | -0.77 (0.157) | -0.55 (0.186)

4. Secondary Outcome: 24h Trough FEV1
Description: Trough FEV1 was defined as the mean of the post-dose 23 h 15 min and the 23 h 45 min FEV1 values. This was measured using central spirometry according to ATS/ERS standardization. This was analyzed using the same MIXED model as specified for the primary analysis.
Time Frame: Day 1, Week 26
Population: The number of participants considered for the analysis was from the full analysis set (randomized participants who received at least one dose of study medication). However, for a given time frame, analyzed participants had values at both baseline and the corresponding time frame, i.e. day 1 or week 26.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | NVA237 | Placebo
Number analyzed (Participants) | 305 | 154
Liters
  Day 1 (n=289,151) | 1.230 (0.0084) | 1.109 (0.0104)
  Week 26 (n=281,143) | 1.195 (0.0140) | 1.059 (0.0171)

5. Secondary Outcome: FEV1 and Forced Vital Capacity (FVC)
Description: FEV1 and FVC were measured using central spirometry according to ATS/ERS standardization. Both were analyzed using the same MIXED model as specified for the primary analysis.
Time Frame: Day 1 at 5, 15, 30 minutes (min) and 1 hour (h) post dose; days 2, 86, 184 at 23 (h) 15 min and 23 h 45 min post dose; days 29, 85, 183 at -45 and -15 min pre-dose and 5, 15, and 30 min post dose
Population: The number of participants considered for the analysis was from the full analysis set (randomized participants who received at least one dose of study medication). However, for a given time frame, analyzed participants had values at both baseline and the corresponding time frame, e.g. day 1, 5 min; day 1, 15 min, etc..
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | NVA237 | Placebo
Number analyzed (Participants) | 305 | 154
Liters
  FEV1, day 1, 5 min (n=281,143) | 1.199 (0.0060) | 1.112 (0.0072)
  FEV1, day 1, 15 min (n=277,147) | 1.245 (0.0075) | 1.116 (0.0089)
  FEV1, day 1, 30 min (n=283,145) | 1.265 (0.0076) | 1.111 (0.0090)
  FEV1, day 1, 1 h (n=284,142) | 1.295 (0.0079) | 1.124 (0.0096)
  FEV1, day 2, 23 h 15 min (n=267,137) | 1.228 (0.0086) | 1.101 (0.0108)
  FEV1, day 2, 23 h 45 min min (n=272,140) | 1.230 (0.0092) | 1.107 (0.0112)
  FEV1, day 29, -45 min (n=273,136) | 1.208 (0.0114) | 1.079 (0.0144)
  FEV1, day 29, -15 min (n=280,142) | 1.226 (0.0113) | 1.097 (0.0142)
  FEV1, day 29, 5 min (n=271,136) | 1.240 (0.0118) | 1.097 (0.0148)
  FEV1, day 29, 15 min (n=272,135) | 1.259 (0.0117) | 1.103 (0.0147)
  FEV1, day 29, 30 min (n=279,139) | 1.272 (0.0114) | 1.105 (0.0142)
  FEV1, day 85, -45 min (n=269,130) | 1.179 (0.0118) | 1.050 (0.0147)
  FEV1, day 85, -15 min (n=271,136) | 1.190 (0.0106) | 1.052 (0.0134)
  FEV1, day 85, 5 min (n=262,130) | 1.229 (0.0119) | 1.059 (0.0147)
  FEV1, day 85, 15 min (n=267,133) | 1.246 (0.0117) | 1.061 (0.0147)
  FEV1, day 85, 30 min (n=273,137) | 1.263 (0.0129) | 1.077 (0.0156)
  FEV1, day 85, 1 h (n=274,133) | 1.275 (0.0125) | 1.079 (0.0154)
  FEV1, day 86, 23 h 15 min (n=261,127) | 1.195 (0.0146) | 1.057 (0.0175)
  FEV1, day 86, 23 h 45 min (n=250,132) | 1.203 (0.0138) | 1.067 (0.0163)
  FEV1, day 183, -45 min (n=262,135) | 1.176 (0.0148) | 1.032 (0.0176)
  FEV1, day 183, - 15 min (n=265,135) | 1.179 (0.0130) | 1.052 (0.0165)
  FEV1, day 183, 5 min (n=262,135) | 1.220 (0.0136) | 1.055 (0.0170)
  FEV1, day 183, 15 min (n=261,140) | 1.233 (0.0139) | 1.070 (0.0169)
  FEV1, day 183, 30 min (n=270,138) | 1.265 (0.0134) | 1.071 (0.0170)
  FEV1, day 183, 1 h (n=263,135) | 1.263 (0.0137) | 1.075 (0.0168)
  FEV1, day 184, 23 h 15 min (n=263,128) | 1.197 (0.0154) | 1.068 (0.0188)
  FEV1, day 184, 23 h 45 min (n=266,132) | 1.196 (0.0144) | 1.058 (0.0180)
  FVC, day 1, 5 min (n=281,143) | 2.925 (0.0184) | 2.739 (0.0220)
  FVC, day 1, 15 min (n=277,147) | 2.992 (0.0252) | 2.759 (0.0288)
  FVC, day 1, 30 min (n=283,145) | 3.041 (0.0235) | 2.761 (0.0280)
  FVC, day 1, 1 h (n=284,142) | 3.044 (0.0240) | 2.755 (0.0286)
  FVC, day 2, 23 h 15 min (n=267,137) | 2.953 (0.0275) | 2.716 (0.0326)
  FVC, day 2, 23 h 45 min (n=272,140) | 2.981 (0.0261) | 2.744 (0.0311)
  FVC, day 29, -45 min (n=273,136) | 2.908 (0.0324) | 2.690 (0.0375)
  FVC, day 29, -15 min (n=280,142) | 2.927 (0.0312) | 2.730 (0.0371)
  FVC, day 29, 5 min (n=271,136) | 2.970 (0.0292) | 2.725 (0.0353)
  FVC, day 29, 15 min (n=272,135) | 2.993 (0.0276) | 2.751 (0.0339)
  FVC, day 29, 30 min (n=279,139) | 2.995 (0.0287) | 2.737 (0.0341)
  FVC, day 85, -45 min (n=269,130) | 2.854 (0.0321) | 2.611 (0.0385)
  FVC, day 85, -15 min (n=271,136) | 2.898 (0.0318) | 2.627 (0.0373)
  FVC, day 85, 5 min (n=262,130) | 2.927 (0.0321) | 2.633 (0.0380)
  FVC, day 85, 15 min (n=267,133) | 2.954 (0.0328) | 2.647 (0.0387)
  FVC, day 85, 30 min (n=273,137) | 2.977 (0.0330) | 2.695 (0.0383)
  FVC, day 85, 1 h (n=274,133) | 2.987 (0.0347) | 2.662 (0.0400)
  FVC, day 86, 23 h 15 min (n=261,127) | 2.908 (0.0366) | 2.612 (0.0429)
  FVC, day 86, 23 h 45 min (n=250,132) | 2.894 (0.0360) | 2.671 (0.0412)
  FVC, day 183, -45 min (n=262,135) | 2.858 (0.0379) | 2.604 (0.0430)
  FVC, day 183, -15 min (n=265,135) | 2.862 (0.0359) | 2.633 (0.0415)
  FVC, day 183, 5 min (n=262,135) | 2.927 (0.0368) | 2.672 (0.0426)
  FVC, day 183, 15 min (n=261,140) | 2.957 (0.0365) | 2.679 (0.0420)
  FVC, day 183, 30 min (n=270,138) | 2.988 (0.0366) | 2.707 (0.0428)
  FVC, day 183, 1 h (n=263,135) | 2.941 (0.0401) | 2.668 (0.0453)
  FVC, day 184, 23 h 15 min (n=263,128) | 2.869 (0.0386) | 2.664 (0.0452)
  FVC, day 184, 23 h 45 min (n=266,132) | 2.894 (0.0402) | 2.647 (0.0472)

6. Secondary Outcome: Peak FEV1
Description: Peak FEV1 was defined as the maximum FEV1 0-4 h post-dose. Peak Fev1 was measured at 45min and 15min pre-dose and up to 4h post dose at day 1, week 12 and week 26, using central spirometry according to ATS/ERS standardization. It was analyzed using the same MIXED model as specified for the primary analysis.
Time Frame: Day 1, week 12, week 26
Population: The number of participants considered for the analysis was from a Serial Spirometry subgroup of the full analysis set where N = 134 and 58, respectively. However, analyzed participants had values at both baseline and the corresponding time frame, i.e. day 1, week 12 or week 26.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | NVA237 | Placebo
Number analyzed (Participants) | 134 | 58
Liters
  Day 1 (n=134,57) | 1.376 (0.0119) | 1.183 (0.0146)
  Week 12 (n=125,56) | 1.347 (0.0207) | 1.140 (0.0245)
  Week 26 (n=124,57) | 1.308 (0.0250) | 1.112 (0.0298)

7. Secondary Outcome: Standardized FEV1 Area Under the Curve (AUC(5 Min-4 h)) Post-dose
Description: The standardized (with respect to time) AUC for FEV1 was calculated between 5 min and 4h post morning dose at day 1, week 12 and week 26. The AUC (5 min-4 h) for FEV1 at each visit was analyzed using the same MIXED model as specified for the primary analysis.
Time Frame: Day 1, week 12, week 26
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | NVA237 | Placebo
Number analyzed (Participants) | 134 | 58
Liters
  Day 1 (n=134,57) | 1.311 (0.0122) | 1.117 (0.0142)
  Week 12 (n=125,56) | 1.286 (0.0204) | 1.080 (0.0241)
  Week 26 (n=124,57) | 1.243 (0.0229) | 1.046 (0.0280)

8. Secondary Outcome: Change From Baseline in Chronic Obstructive Pulmonary Disease (COPD) Symptoms (Cough, Wheezing, Shortness of Breath, Sputum Volume, Sputum Color and Night Time Awakenings)
Description: In an electronic diary, the participant responded to 6 questions twice daily to report on the degree of symptoms over the past 12 hours of the morning and evening. The questions covered the participant's degree of overall symptoms, and degrees of individual symptoms of coughing, wheezing, amount of sputum, color of sputum and breathlessness. Each question scored from 0 to 3 where 0 represented no symptom present and 3 represented the worst degree of that symptom. A negative change in symptom score indicates improvement.
Time Frame: Baseline, 26 weeks
Population: The number of participants considered for the analysis was from the full analysis set (randomized participants who received at least one dose of study medication). However, for a given symptom category, analyzed participants had both baseline and week 26 values.
Measure: Least Squares Mean (Standard Error); unit: score
Arm/Group | NVA237 | Placebo
Number analyzed (Participants) | 305 | 154
score
  Total symptom (n=296,150) | -1.16 (0.143) | -0.85 (0.164)
  Respiratory symptom | -0.21 (0.033) | -0.12 (0.038)
  Cough symptom | -0.24 (0.030) | -0.20 (0.036)
  Wheeze symptom | -0.30 (0.030) | -0.22 (0.036)
  Sputum production | -0.15 (0.034) | -0.11 (0.039)
  Sputum color | -0.10 (0.025) | -0.10 (0.031)
  Breathless symptom | -0.17 (0.030) | -0.10 (0.035)

9. Secondary Outcome: Time to First Moderate or Severe COPD Exacerbation
Description: A COPD exacerbation was defined as a worsening of the following two or more major symptoms for at least 2 consecutive days:1) dyspnea; 2) sputum volume; 3) sputum purulence; or defined as a worsening of any 1 major symptom together with an increase in any 1 of the following minor symptoms for at least 2 consecutive days: 1) sore throat; 2) colds (nasal discharge and/or nasal congestion); 3) fever without other cause; 4) cough; 5) wheeze. COPD exacerbations were recorded in the patient diary and other source documents.
Time Frame: 26 weeks
Population: Full Analysis Set: The full analysis set included all randomized patients who received at least one dose of study medication.
Measure: Median (Full Range); unit: Days
Arm/Group | NVA237 | Placebo
Number analyzed (Participants) | 305 | 154
Days | NA [NA to NA] — The median time was not estimable due to the low number of participants with moderate or severe COPD exacerbations. | NA [NA to NA] — The median time was not estimable due to the low number of participants with moderate or severe COPD exacerbations.

10. Secondary Outcome: Number of Moderate and Severe COPD Exacerbations
Description: COPD exacerbations were recorded in the patient diary and other source documents. The rate of COPD exacerbations during the 26 week treatment period was analyzed using a generalized linear model assuming a negative binomial distribution.
Time Frame: 26 weeks
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Number of exacerbations
Arm/Group | NVA237 | Placebo
Number analyzed (Participants) | 305 | 154
Number of exacerbations | 0.2 (0.48) | 0.3 (0.58)

11. Secondary Outcome: The Total Score of the St George's Respiratory Questionnaire (SGRQ)
Description: SGRQ is a health related quality of life questionnaire consisting of 51 items in three components: symptoms, activity and impacts. The lowest possible score is zero and the highest possible score is 100. Higher scores correspond to greater impairment in quality of life. The health-related quality of life was measured using SGRQ. It was completed by the participant at the investigators site.
Time Frame: Week 12, week 26
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Score
Arm/Group | NVA237 | Placebo
Number analyzed (Participants) | 305 | 154
Score
  week 12 (n=293,147) | 32.35 (1.232) | 37.39 (1.399)
  week 26 (n=288,144) | 31.02 (1.480) | 35.94 (1.641)

ADVERSE EVENTS:
Arm/Group | NVA237 | Placebo
Serious Adverse Events (participants affected / at risk) | 17/305 | 14/154
Other Adverse Events (participants affected / at risk) | 81/305 | 48/154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NVA237 (N=305) | Placebo (N=154)
Angina pectoris (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cor pulmonale chronic (Cardiac disorders) | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Death (General disorders) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 2 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 3
Viral infection (Infections and infestations) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 2 | 0
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral arteriosclerosis (Nervous system disorders) | 1 | 0
Thalamus haemorrhage (Nervous system disorders) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 10 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Shock (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NVA237 (N=305) | Placebo (N=154)
Nasopharyngitis (Infections and infestations) | 36 | 15
Upper respiratory tract infection (Infections and infestations) | 18 | 12
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 49 | 32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.